CLINICAL TRIAL: NCT04430673
Title: VR4REHAB-MOTIVATION for REHABILITATION: Proof of Concept Evaluation of Virtual Reality Innovations for Therapy for Young People With Brain Injury
Brief Title: Virtual Rehabilitation Innovations for Motivation
Acronym: VR4REHAB-MOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Free Hospital NHS Foundation Trust (Other)
Collaborators: Interreg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRAS 275096
Record Dates: First submitted 2020-04-22; First posted 2020-06-12 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Virtual Rehabilitation; CP (Cerebral Palsy); Brain Injuries; Young Adult; Children
Keywords: Virtual Rehabilitation; Cerebral palsy; Acquired brain injury; children and young people
MeSH Terms: conditions — Cerebral Palsy; Brain Injuries

STUDY DESIGN:
Intervention Model Description: Action Research Proof of Concept study in 2-Phases. Phase 1, 2-hour workshop: Phase 2 2-week within subject trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home-School based VR trial (Experimental): The VR system will be provided to each participant for a 2-week home- or school- based trial. No additional interventions.
  Interventions: Other: Home-School based VR system trial

INTERVENTIONS:
Other: Home-School based VR system trial — Commercially available VR games operated Raspberry pi micro computer and Oculus Quest VR headsets provided for 2 weeks at dose and intensity selected by participants.

SUMMARY:
Children and young people with movement difficulties such as Cerebral Palsy (CP) and Acquired Brain Injury (ABI) report that traditional therapies are highly repetitive and labourious. This influences enjoyment and participation in regular therapy programmes and may result in reduced adherence to therapy or exercise regimes, limiting effectiveness. This study will build on the team's previous work to explore the potential use of Virtual-Reality (VR) technologies in rehabilitation; particularly systems that can be used at home to increase accessibility and reduce need to attend clinics for therapy. During the co-production events of the VR4REHAB Inter Regional North West Europe (NWE) funded programme in 2018, young people desired the use of commercial games for therapeutic purposes. This work has enabled connections between affordable computer technologies: the Raspberry Pi, VR headsets and freely available commercial games.

This 2-Phased project is therefore exploring the potential of commercially available virtual reality (VR) systems consoles and games for use in rehabilitation programmes. The Investigators hope to gain information on:

1. Whether commercially produced VR games can provide a motivating environment to support adherence to therapy
2. Whether it is possible to improve reaching and grasp-release hand movements through this method
3. Gain an understanding of the ages of children and young people most likely to benefit from home-based VR therapy User evaluation and performance data and therapist evaluations will be collected and compared to baseline data to provide information on usability, accessibility, acceptability and adaptability.

DETAILED DESCRIPTION:
Aim: The focus of this Proof-of-Concept feasibility study investigates the potential of commercially available virtual reality (VR) games and equipment for therapeutic use for upper limb rehabilitation; considering in particular the role of motivation and engagement when using the system to support adherence to therapy protocols.

Rationale - Effective rehabilitation requires appropriate dosage and intensity and be meaningful to daily life, but traditional therapeutic modalities struggle to achieve optimum input and gains following successful intensive intervention programmes are often not maintained. Commercial VR products are designed with high level gaming methods to engage participants in the games. Commercial VR products therefore offer potential as therapeutic adjuncts to gain appropriate practice of sufficient intensity and duration but may need some adjustments. Adjustments in this instance refer to changing the speed at which the game plays and which combinations of devices compliant with European Union standards (CE) can be connected.

The Investigators will evaluate whether young people with Cerebral Palsy (CP) or Acquired Brain injury (ABI) can be engaged in VR games for upper-limb movement using VR systems, potential for therapeutic benefit and also consider clinical feasibility in relation to utility, particularly in respect to the costs involved (i.e. labour, training, workplace set-up). The Co-Production Group (C-PG) group identified a 2-Phase study in order to assess for any modifiable alterations and prepare training manual prior to a short feasibility trial. This clinical trial is designed as an Action Research study in two Phases:

Phase 1 of the study. Participants will engage in a 2-hour workshop to test out the VR system and games in order to gather responses to the game speeds and devices (including method of access). Feedback will contribute to information for instruction leaflets for access and usability and determine whether further adjustments are required and additional training information needed for therapists to be able to set up the system to meet individual requirements. Information gathered during the workshop will also inform on the links and support required from the computer scientists for backup.

Phase 2 of the study, will test out the feasibility of use within a home/school setting as a Proof-of-Concept study. Phase 2, will inform on trial design for a larger randomized controlled trial. The VR system will be provided to each participant for a 2-week home- or school- based trial. User evaluation and performance data and therapist evaluations will be collected and compared to baseline data to provide information on usability, accessibility, acceptability and adaptability.

Evidence from preliminary, albeit small single-subject design studies, suggests that children and adults with movement impairments may improve upper limb performance (speed, fluency and accuracy) with some transfer to clinical measures of upper limb and hand skills. It is not known if children with CP/ABI can improve upper limb movement performance and function nor whether gains transfer into improved hand skills in daily life although it anticipated that benefits to function will be achieved for many children. An exploration of this point will be considered as secondary outcomes to inform on dose and duration for a future definitive clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Bilateral and Unilateral CP or ABI with movement difficulties; Gross Motor Function Classification System (GMFCS) levels I to IV e.g. able to sit, independently operate electric wheelchair;
2. Manual Ability Classification System (MACS) levels I to IV - able to move arms and hands and interact with some objects although adaptations may be needed to hold console/interfacing device such as use of velcro strap;
3. Ability to follow simple task instruction;
4. Aged 10 - 30 years; 5)) Ability to cooperate with assessment instructions.

6) Ability to give informed consent or assent if appropriate, participants having an acceptable individual capable of giving consent on the participant's behalf (e.g. parent or guardian of a child under 16 years of age)

* Typically developed peers will need to meet criteria 3 to 6 and be eligible with respect to exclusion criteria.

Exclusion Criteria:

1. Individuals who are GMFCS or MACS levels V; Inability to follow simple task instructions;
2. less than 10 years or over 30 years;
3. Individual with photosensitive epilepsy
4. Unstable medical condition (in -patient status)
5. Learning or behavior difficulties limiting ability to follow instructions or attend a 2 hour workshop/engage with a rehabilitation programme.
6. Receiving Motor therapy treatment (eg. Botulinum Toxin Injections/A/Constraint Induced Movement Therapy or anticipated to receive such treatment during the 6 months of the study

Ages: 10 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
User Evaluation Questionnaire Form | Phase 2: 2-weeks (end of 2-week trial)
  User evaluation (experience) questionnaire developed by the Co-production group. 15 closed questions rate aspects of accessibility and usability, enjoyment and relatedness and 5 open-ended questions for more personal feedback of experience, potential for use in rehabilitation and any recommended changes. Total scores will be computed with descriptive statistics recorded. Content and thematic analysis will be used to analyse data from open ended questions and considered with respect to the ratings provided by participants.
Participant completed engagement diary | Phase 2: Daily over 2 weeks
  Diaries of participants in which they note whether they chose or were prompted to use the game/system and record their experience of the session along with numbers of games played and reported duration of the session. Qualitative methods using content and thematic analysis will be used to analyse data to assist understanding of barriers or facilitators to user engagement.

SECONDARY OUTCOMES:
Goal Attainment Scaling | Phase 2: Day 1 and at 2-weeks (end of 2-week trial)
  Patient reported outcomes using Goal Attainment Scaling will consider potential of system to address 3 identified child/young adult identified goals. Anticipated outcomes are defined on a 5 point scale with -2 = a much less than anticipated outcome; -1= less than anticipated outcome; 0=anticipated outcome; +1 =better than expected outcome; +2=much better than expected outcome. Each goal is weighted by asking the participant to rank them in order of importance and also with respect to anticipated difficulty on a four point scale and a total weigh/per goal determined by multiplying Importance x difficulty=weight of goal. The outcome score for each goal is rated at the review data and the goal attainment 'T-score' calculated using the formula and calculation provided in Turner Stokes (2006) which takes into consideration the sum of weights and score changes and expected correlations. HIgher scores reflect better outcome.
Functional Reach Test | Phase 2: Day 1 and at 2-weeks (end of 2-week trial)
  Functional Reach test measures extent of forward reach of each arm in centimetres while maintaining balance. Larger distance is better function.

OTHER OUTCOMES:
Therapist diary of experiences | Phase 2: Daily over 2 weeks
  Research therapists will record the type of support provided to participants, training requirements and their opinion as to whether the system supported therapeutic objectives in order to consider feasibility of delivery. Comments will be analysed qualitatively to understand the types of support and/or refinements to the system set up or information required for participants to use the system at home.
Therapist diary of time | Phase 2: Daily over 2 weeks
  Research therapists and level of experience/salary banding will record the amount of time provided to participants and any additional training time. Total time will be calculated to determine potential cost to support home-based use of VR systems.

CONTACTS AND LOCATIONS:
Overall Officials: Research and Development Manager, Study Chair — Research Sponsor
Locations (1):
- Royal Free London NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
This is a small study involving qualitative feedback and releasing individual data would risk contributing to misleading interpretations if added to a larger data set.